CLINICAL TRIAL: NCT05025267
Title: Prospective Study of Ability to Meet Nutritional Needs with a Peptide-based, High Protein Enteral Formula
Brief Title: Ability to Meet Enteral Nutritional Needs with a Peptide-based, High Protein Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19.01.CA.HCN
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Enteral Feeding

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, non-randomized, open-label observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enteral Tube-fed Adults (Other): Adults being fed an enteral formula with a feeding tube
  Interventions: Other: Medical Food: Peptide-Based Enteral Formula

INTERVENTIONS:
Other: Medical Food: Peptide-Based Enteral Formula — Will be fed exclusively the study peptide-based, high protein enteral formula via a feeding tube

SUMMARY:
This is a prospective, open-label single-arm observational clinical trial to assess enteral feeding nutrition goals with a peptide-based, high protein enteral formula.

DETAILED DESCRIPTION:
This is a prospective, observational study to assess the ability to meet enteral nutrition goals and tolerance of a peptide-based, high protein tube feeding product in adult, tube-fed patients living in the community setting. In addition, the study will explore metabolic and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Adults with established enteral access
* Anticipated to require enteral nutrition to provide 90% or more of their nutritional needs
* Signed informed consent

Exclusion Criteria:

* Condition which contraindicates enteral feeding (i.e. intestinal obstruction)
* Any condition that would contraindicate use of the study product
* Patients with active colitis, radiation enteritis, SBS, undergoing active cancer treatment
* Judged to be at risk for poor compliance to the study protocol
* Participating in a conflicting clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Calorie nutritional goals | 14 days
  Daily percentage of calorie nutritional goals met

SECONDARY OUTCOMES:
Protein nutritional goals | 14 days
  Daily percentage of protein nutritional goals met
Daily reports of gastrointestinal intolerance | 14 days
  Daily occurrence of nausea, stool frequency, stool consistency, and/or vomiting)
Adverse events | 14 days
  Daily adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Krysmaru Araujo Torres, MD, Study Director — Nestle Health Science
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No